CLINICAL TRIAL: NCT00907439
Title: Changes in Diastolic Dysfunction With the Onset of Volatile Anesthesia in Patients Undergoing Coronary Artery Bypass Grafting as Determined by a Load-independent Efficiency Index Derived From the Parameterized Doppler Analysis of Left Ventricular Filling
Brief Title: Study of the Effect of Inhaled Anesthetics on Diastolic Heart Function Using a Doppler-derived Efficiency Index
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Troy Wildes, MD, Assistant Professor, Washington University School of Medicine, Department of Anesthesiology
Other Study IDs: WU-HRPO-07-0551
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-11

CONDITIONS: Diastolic Dysfunction; Coronary Artery Disease; General Anesthesia
Keywords: Diastole, physiopathology; coronary artery disease; volatile anesthetic; sevoflurane
MeSH Terms: conditions — Coronary Artery Disease; Heart Murmurs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the effect of inhaled anesthetic drugs upon diastolic heart function (heart suction and filling performance) in patients who are undergoing coronary bypass surgery.

DETAILED DESCRIPTION:
Diastolic heart dysfunction is a significant cause of cardiovascular morbidity and is the cause of symptomatic heart failure in approximately one half of patients who are admitted to hospitals with heart failure symptoms. However, diastolic heart function remains difficult to measure objectively without cardiac catheterization. Diastolic heart dysfunction is also common among patients undergoing coronary bypass grafting (CABG) surgery. Despite the ubiquitous use of inhaled volatile drugs to maintain anesthesia in these patients, their effects upon diastolic heart function remain unclear.

ELIGIBILITY:
Inclusion Criteria:

* Non-emergent coronary bypass grafting surgery
* Left ventricular ejection fraction of 40% or greater

Exclusion Criteria:

* Myocardial infarction within 4 weeks
* Greater than mild cardiac valvular pathology
* Body mass index greater than 35
* Cardiac dysrhythmias or pacemaker therapy
* Left bundle branch block
* Uncontrolled gastroesophageal reflux disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing non-emergent coronary artery bypass grafting surgery at a tertiary care center
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Diastolic efficiency index (derived from the parameterized analysis of transmitral early filling Doppler using the paradigm of the ventricle as a damped harmonic oscillator) | Following induction of volatile anesthesia

SECONDARY OUTCOMES:
Diastolic efficiency index (derived from the parameterized analysis of transmitral early filling Doppler using the paradigm of the ventricle as a damped harmonic oscillator) | Following the onset of controlled ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Troy S Wildes, MD, Principal Investigator — Washington University School of Medicine, Department of Anesthesiology
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Shmuylovich L, Kovacs SJ. Load-independent index of diastolic filling: model-based derivation with in vivo validation in control and diastolic dysfunction subjects. J Appl Physiol (1985). 2006 Jul;101(1):92-101. doi: 10.1152/japplphysiol.01305.2005. Epub 2006 Mar 30. PMID 16575023
- [Background] Boskovski MT, Shmuylovich L, Kovacs SJ. Transmitral flow velocity-contour variation after premature ventricular contractions: a novel test of the load-independent index of diastolic filling. Ultrasound Med Biol. 2008 Dec;34(12):1901-8. doi: 10.1016/j.ultrasmedbio.2008.05.002. Epub 2008 Aug 9. PMID 18692298